CLINICAL TRIAL: NCT02098473
Title: A Phase2, Multi-Center, Multi-national, Randomized, Double-blind, Placebo-controlled Parallel-group Clinical Trial to Evaluate the Efficacy and Safety of RPC4046 in Adult Subjects With Eosinophilic Esophagitis
Brief Title: Dose Ranging Study of RPC4046 in Eosinophilic Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPC02-201
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — cendakimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- RPC4046 Low Dose (Experimental): intravenous (IV) infusion only once at first dose, 2 subcutaneous (SC) injections weekly for 16 weeks, low dose
  Interventions: Drug: RPC4046
- RPC4046 High Dose (Experimental): intravenous (IV) infusion only once at first dose, 2 subcutaneous (SC) injections weekly for 16 weeks, high dose
  Interventions: Drug: RPC4046
- Placebo (Placebo Comparator): intravenous (IV) infusion only once at first dose, 2 subcutaneous (SC) injections weekly for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RPC4046
  Arms: RPC4046 High Dose; RPC4046 Low Dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effective dose(s) of RPC4046 in the treatment of Eosinophilic Esophagitis (EoE). This trial consists of two phases: 16 weeks of double-blind treatment and 52 weeks of open-label extension.

ELIGIBILITY:
Inclusion Criteria:

* Histologic evidence of EoE
* Clinical symptoms of EoE including dysphagia

Exclusion Criteria:

* Primary causes of esophageal eosinophilia other than EoE

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08-31 (Actual); Primary Completion 2016-02-17 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Mean Eosinophil Count | Week 16

CONTACTS AND LOCATIONS:
Locations (30):
- United States (27):
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - Desert Sun Clinical Research, LLC, Tucson, Arizona
  - Alliance Clinical Research, Oceanside, California
  - Precision Research Institute, LLC, San Diego, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - University of Florida, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Children's Center for Digestive Healthcare, Atlanta, Georgia
  - Grand Teton Research Group, Idaho Falls, Idaho
  - Northwestern University-Feinberg School of Medicine, Chicago, Illinois
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Gastroenterology and Hepatology Service Walter Reed National Military Medical Center, Bethesda, Maryland
  - Metropolitan Gastroenterology Group Chevy Chase Clinical Research, Chevy Chase, Maryland
  - West Michigan Clinical Research Center Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - Minnesota Gastroenterology, Plymouth, Minnesota
  - GI Associates and Endoscopy Center-GI Clinical Research Department, Flowood, Mississippi
  - Darthmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Great Lakes Gastroenterology Research, Mentor, Ohio
  - University of Pennsylvania Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Utah Division of Gastroenterology, Salt Lake City, Utah
- Gastrointestinal Research Group, University of Calgary Health, Calgary, Alberta, Canada
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Swiss EoE Clinic, Olten

REFERENCES:
- [Derived] Caldwell JM, Ballaban AY, Li J, Maddux R, Harris S, Dellon ES, Rothenberg ME. Cendakimab (anti-IL-13) administration improves esophageal gene expression in eosinophilic esophagitis. J Allergy Clin Immunol. 2026 Jan;157(1):118-130.e7. doi: 10.1016/j.jaci.2025.08.032. Epub 2025 Oct 9. PMID 41067281
- [Derived] Dellon ES, Collins MH, Rothenberg ME, Assouline-Dayan Y, Evans L, Gupta S, Schoepfer A, Straumann A, Safroneeva E, Rodriguez C, Minton N, Hua SY, Hirano I. Long-term Efficacy and Tolerability of RPC4046 in an Open-Label Extension Trial of Patients With Eosinophilic Esophagitis. Clin Gastroenterol Hepatol. 2021 Mar;19(3):473-483.e17. doi: 10.1016/j.cgh.2020.03.036. Epub 2020 Mar 21. PMID 32205221
- [Derived] Hirano I, Collins MH, Assouline-Dayan Y, Evans L, Gupta S, Schoepfer AM, Straumann A, Safroneeva E, Grimm M, Smith H, Tompkins CA, Woo A, Peach R, Frohna P, Gujrathi S, Penenberg DN, Li C, Opiteck GJ, Olson A, Aranda R, Rothenberg ME, Dellon ES; HEROES Study Group. RPC4046, a Monoclonal Antibody Against IL13, Reduces Histologic and Endoscopic Activity in Patients With Eosinophilic Esophagitis. Gastroenterology. 2019 Feb;156(3):592-603.e10. doi: 10.1053/j.gastro.2018.10.051. Epub 2018 Nov 2. PMID 30395812